CLINICAL TRIAL: NCT02071212
Title: A Single Center Phase II Assessor-Blinded RaNdomised Active Controlled Parallel-Group Trial to COmpare Ticagrelor Versus Clopidogrel on the REduction of ArteriaL STiffness and Wave Reflections in Patients With CoronarY Artery Disease.
Brief Title: Compare Ticagrelor vs Clopidogrel on the Reduction of Arterial Stiffness and Wave Reflectionsin Patients With CAD.
Acronym: NOVELTY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Cardiovascular Research Society (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D5130L00063
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel (Active Comparator): Loading dose 600 mg .Mainatinance dose 75 mg QD
  Interventions: Drug: Ticagrelor
- Ticagrelor (Experimental): Loading dose 180 mg . Maintenance 90 mg BID
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Loading dose 180 mg . Maintainance dose 90 mg BID
  Other Names: BRILIQUE

SUMMARY:
The purpose of this study is to investigate the potential acute and chronic effect of ticagrelor versus clopidogrel on arterial stiffness and other vascular risk markers of interest, the study will consist of two periods: a 24-hour ACUTE period where 60 subjects with an indication for coronary angiography (CA) with or without percutaneous coronary intervention (PCI) will be included, and a 30-day CHRONIC period where approximately 60 subjects that will undergo PCI will be included and studied (refer to Section 3 'Study Plan and Procedures'). The primary objective of this study is to compare ticagrelor versus clopidogrel regarding their effect on arterial stiffness as assessed by PWV, at 3 hours after the loading dose of each regimen, in eligible subjects with CAD.

DETAILED DESCRIPTION:
This is singe-center, randomized, assessor-blinded, active controlled, parallel-group trial consisting of an 'acute' and a 'chronic' period, aiming at comparing ticagrelor versus clopidogrel on the reduction of arterial stiffness and wave reflections in patients with CAD. This Investigator-Sponsored Study (ISS) will be supported by AstraZeneca.

60 subjects fulfilling all study-specific eligibility criteria will be initially recruited for the 'acute' study period of 24-hour duration. Subjects that will undergo ad hoc PCI will continue in the subsequent 'chronic' study period of 30-day duration.

In order to have 60 subjects in the 'chronic' study period (since some of the 'acute' period will not undergo PCI), additional subjects that are scheduled for elective PCI will be recruited until the sample size of 'chronic' study period reaches 60 subjects.

The study periods [Figure 1, Flow Chart] have as follows:

For the 24-hour ACUTE period, 60 subjects with an indication for elective CA with or without PCI will be included in the study.

Three (3) hours before the CA the subjects will be randomized in the two study treatment arms:

Ticagrelor arm: 30 subjects will receive

* 180 mg loading dose of ticagrelor,
* 1st maintenance ticagrelor dose of 90 mg at 12 hours. Clopidogrel arm: 30 subjects will receive
* 600 mg loading dose of clopidogrel.

Study measurements (arterial stiffness, central blood pressure and endothelial function) for both study treatment arms will be performed at:

* baseline (0 hours - prior to the loading dose administration)
* 3 hours (after the loading dose of each regimen and before CA), and at
* 24 hours (before the administration of the 2nd maintenance dose of ticagrelor and the 1st maintenance dose of clopidogrel).

For the 30-day CHRONIC period, 60 subjects that will undergo PCI (stent implantation) will be studied. Part of this 'chronic' period population will consist of the subjects that were included in the 'acute' period and proceeded ad hoc to PCI. The remainder will be subjects being scheduled for elective PCI, who will be enrolled after the completion of the recruitment in the 'acute' study period.

Approximately 30 subjects will be allocated to ticagrelor loading dose and maintenance dose (90 mg BID) thereafter and approximately 30 subjects will be allocated to 600 mg of clopidogrel and maintenance dose (75 mg QD) thereafter.

Study measurements for the subjects of the 'acute' period that will enter the 'chronic' period will be performed at:

- 30 days post-PCI (prior to the administration of the morning maintenance dose of the assigned treatment regimen at the day of study visit).

Study measurements for the additional subjects with indication of elective PCI that will be enrolled directly into the chronic study period will be performed at:

* baseline (0 hours - prior to the administration of the loading dose of each treatment regimen and 3 hours before the PCI)
* 30 days post PCI (prior to the administration of the morning maintenance dose of the assigned treatment regimen at the day of study visit).

All study-related procedures will be carried out in accordance with the institutional guidelines and common practice.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Male and female subjects > 18 and < 79 years of age.
3. Indication for elective coronary angiography (angina, positive stress test/SPECT/stress echo) with or without PCI for inclusion in the 'acute' study period, and indication for either ad hoc or elective PCI for inclusion in the 'chronic' study period.

Exclusion Criteria:

1. Who had ACS within 12 months of screening.
2. Previous stent implantation with dual antiplatelet therapy within 12 months of screening.
3. Subjects being treated with anti-platelet medications other than aspirin prior to diagnostic catheterization including glycoprotein IIb/IIIa inhibitors.
4. Subjects with NYHA class III or IV heart failure or known left ventricular ejection fraction < 30%.
5. Subjects with hemodynamic or electrical instability (including shock).
6. History of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 6 months.
7. Other bleeding diathesis, or considered by Investigator to be at high risk for bleeding.
8. Any previous history of ischemic or hemorrhagic stroke, intracranial hemorrhage or disease (neoplasm, arteriovenous malformation, aneurysm).
9. International Normalized Ratio (INR) known to be >1.5 within 1 week of study entry.
10. Poorly controlled blood pressure (>160/100 mmHg).
11. Known platelet count of <100,000/mm3 within 1 week of study entry.
12. Known anemia (hemoglobin [Hb] <10 gr/dL) within 1 week of study entry.
13. Subjects receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase-2 (COX-2) inhibitors that cannot be discontinued for the duration of the study.
14. Severe kidney disease (GFR<30 ml/min/1.73m2).
15. Hepatic insufficiency defined as liver cirrhosis, AST/ALT/Alkaline Phosphatase greater than 3 times the upper limit of normal or hyperbilirubinemia defined as peak total serum bilirubin greater than 2 times the upper limit of normal (ULN).
16. Any indication (atrial fibrillation, mitral stenosis or prosthetic heart valve, pulmonary embolism (PE), deep vein thrombosis (DVT)) for anticoagulation treatment during study period.
17. Asthma or chronic obstructive pulmonary disease requiring brochodilating agents.
18. Concomitant use of potent Cytochrome P450 3A4 (CYP3A4) inhibitors (atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin and voriconazole) or inducers (carbamazepine, dexamethasone, phenobarbital, phenytoin, rifampin, and rifapentine).
19. Concomitant use of drugs that are metabolized through CYP2C19 (omeprazole and esomeprazole, fluvoxamine, fluoxetine, moclobemide, voriconazole, fluconazole, ticlopidine, ciprofloxacin, cimetidine, carbamazepine, oxcarbazepine and chloramphenicol).
20. History of uric acid nephropathy and high levels of uric acid within 1 week of study entry.
21. Increased risk of bradycardic events (e.g. known sick sinus syndrome or third degree AV block or previous documented syncope suspected to be due to bradycardia unless treated with a pacemaker).
22. Known neoplastic or autoimmune disease or any concomitant medical illness that in the opinion of the Investigator may interfere with or prevent completion in this study.
23. Contraindication to clopidogrel, ASA, or ticagrelor.
24. A history of alcohol and/or substance abuse that could interfere with conduct of the trial.
25. Pregnancy or lactation (for premenopausal women 2 methods of reliable contraception, one of which must be barrier method, are required).
26. Treatment with other investigational agents (including placebo) or devices within 30 days prior to randomization or planned use of investigational agents or devices prior to the Day 30 visit.
27. Life expectancy less than 1 year.
28. Indication for major surgery (e.g. cancer treatment, carotid surgery, cerebral surgery, major vascular surgery).
29. High likelihood of being unavailable for the Day 30 follow up.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-02; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Mean Change in the cfPWV | at 3 hours after the loading dose
  The primary outcome is the treatment difference in the mean change in cfPWV from baseline (0 hours) at 3 hours after the loading dose of each regimen, in ticagrelor and clopidogrel acute period populations.

SECONDARY OUTCOMES:
mean change in the cfPWV | from baseline at 24 hours after the loading dose
  The treatment difference in the mean change in the cfPWV from baseline (0 hours) at 24 hours after the loading dose of each regimen, in the acute period populations;

CONTACTS AND LOCATIONS:
Overall Officials: Charalambos Vlachopoulos, Principal Investigator — Ippokratio Hospital Athens , Greece
Locations (1):
- Ippokratio Hospital, Athens, Greece

REFERENCES:
- [Derived] Vlachopoulos C, Georgakopoulos C, Pietri P, Ioakeimidis N, Koutouzis M, Vaina S, Aznaouridis K, Toutouzas K, Latsios G, Terentes-Printzios D, Rigatou A, Tousoulis D. Effect of Ticagrelor Versus Clopidogrel on Aortic Stiffness in Patients With Coronary Artery Disease. J Am Heart Assoc. 2019 Jun 18;8(12):e012521. doi: 10.1161/JAHA.119.012521. Epub 2019 Jun 5. PMID 31165663